CLINICAL TRIAL: NCT01909154
Title: Phase I Pilot Study to Evaluate the Security of Local Administration of Autologous Stem Cells Obtained From the Bone Marrow Stroma, in Traumatic Injuries of the Spinal Cord
Brief Title: Safety Study of Local Administration of Autologous Bone Marrow Stromal Cells in Chronic Paraplegia
Acronym: CME-LEM1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Jesús Vaquero Crespo, M.D., Doctor on neurosurgery, Puerta de Hierro University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CME-LEM1; 2010-023285-46 (EudraCT Number)
Record Dates: First submitted 2013-07-07; First posted 2013-07-26 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Spinal Cord Injury
Keywords: neurophysiological parameters improvement; spinal cord injury; biology therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mesenchymal stromal cell therapy (Experimental): Autologous bone marrow adult mesenchymal stem cells expanded in vitro. Administered by Intrathecal injection (subarachnoid and intramedullary). Depending on centromedullary post-traumatic injury: bone marrow stromal stem cells administration (MSCs) at the minimum dose of 100x106 followed by subarachnoid administration of 30x106 MSCs,3 months later
  Interventions: Biological: Mesenchymal stromal cell therapy

INTERVENTIONS:
Biological: Mesenchymal stromal cell therapy — Stem cells administration locally
  Other Names: BMMSCs= Bone Marrow Mesenchymal Stem Cells

SUMMARY:
The purpose of this study is to confirm the security, and detect the effect of the local administration in damaged nervous tissue, of autologous bone marrow stromal cells.

DETAILED DESCRIPTION:
It is a clinical trial phase I, single center, non-randomized, uncontrolled, open prospective follow-up of a cohort of patients with chronic spinal cord injury (SCI) who were treated with autologous stromal cells of the bone marrow administrated locally (subarachnoid and intramedullar) by intrathecal microinjection and three months later, by lumbar subarachnoid administration. The minimum follow-up duration for each patient is 12 months after the first administration, or until death, if it occurs it before.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with ages between 18 years and 60 years with of age or older functional sequelae chronically established by traumatic injury of the spinal cord (spinal segments between the vertebral bodies C6 and L1) and considered irreversible (not respond to any other treatment). In this study, the lesion is considered chronically established, when there are no signs of functional recovery after a minimum follow-up period of 6 months after the spinal cord injury. The upper age limit is justified by the low potential of in vitro expansion of bone marrow stromal cells over 60 years.
* Complete paraplegia, with loss of motor and sensory function below the lesion (grade A in the American Spinal Injury Association Impairment (ASIA) Scale .
* Spinal injury MRI morphologically visible, and without images that suggest spinal cord transection, with separation of the both ends of the spinal cord.
* Tracking evolutionary possibility after treatment protocol and to comply physiotherapy maintained throughout the follow up period.
* Written informed Consent according to good clinical practice (GCP) and local regulations, obtained before any study procedure.
* Hematological parameters and creatinine, serum glutamate oxaloacetate transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) in normal range according to laboratory standards, are accepted, however, small non-significant deviations according to the investigator.

Exclusion criteria:

* Pregnancy and lactation
* Systemic disease represents an added risk to treatment
* Patients with questions about their possible cooperation in rehabilitation-physiotherapy treatments later, or negative report psychological assessment prior.
* Neuroimaging data showing spinal cord section with separation of the terminal portion of the spinal cord
* Current neoplastic disease diagnosed or treated in the previous five years
* Patients treated with hematopoietic growth factors or requiring stable anticoagulation
* Added neurodegenerative disease
* History of substance abuse, psychiatric illness or allergy to protein products used in the process of cell expansion
* HIV positive serology and syphilis
* Hepatitis B or Hepatitis C active According to the investigator's opinion if there are findings on physical examination, abnormal clinical test results or other medica relevant entries, social or psychosocial factors which might influence negatively the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus JV Vaquero Crespo, Dr., Principal Investigator — Hospital Universitario Puerta de Hierro-Majadahonda
Locations (1):
- Hospital Puerta de Hierro, Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
nonymized individual data of participants will be shared with Authorities at the end of the Clinical Development Plan by the CTD (Common Technical Document). Results will be published in a scientific publication.

REFERENCES:
- [Background] Geffner LF, Santacruz P, Izurieta M, Flor L, Maldonado B, Auad AH, Montenegro X, Gonzalez R, Silva F. Administration of autologous bone marrow stem cells into spinal cord injury patients via multiple routes is safe and improves their quality of life: comprehensive case studies. Cell Transplant. 2008;17(12):1277-93. doi: 10.3727/096368908787648074. PMID 19364066

RESULTS

PARTICIPANT FLOW:
Groups:
- Mesenchymal Stromal Cell Therapy: Autologous bone marrow adult mesenchymal stem cells expanded in vitro. Administered by Intrathecal injection (subarachnoid and intramedullary). Depending on centromedullary post-traumatic injury: bone marrow stromal stem cells administration (MSCs) at the minimum dose of 100x10^6 followed by subarachnoid administration of 30x10^6 MSCs,3 months later
  Mesenchymal stromal cell therapy
Period: Overall Study
Arm/Group | Mesenchymal Stromal Cell Therapy
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mesenchymal Stromal Cell Therapy
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  Spain | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety-Number of Adverse Events
Description: Clinical evaluation of possible adverse effects is performed daily at the first week after the first administration of stem cells and weekly until the 6 months follow-up visit and then at month 9 and 12. .
  * During the first stem cells administration (during surgery): Changes in vital signs (ECG, Blood Pressure (BP), Heart Rate (HR) were evaluated
  * During the second stem cells administration: Changes in vital signs (BP, HR), headache and meningeal irritation were evaluated
  * During the first weeks, after the first and the second administrations, the possibility of meningeal irritation, headache and infectious complications were considerate.
  MedDRA stardards are followed
Time Frame: Up to 12 months
Population: Autologous bone marrow adult mesenchymal stem cells expanded in vitro. Administered by Intrathecal injection (subarachnoid and intramedullary). Depending on centromedullary post-traumatic injury: bone marrow stromal stem cells administration (MSCs) at the minimum dose of 100x106 followed by subarachnoid administration of 30x106 MSCs,3 months later
Measure: Number; unit: Adverse events
Groups:
- Mesenchymal Stromal Cell Therapy: Autologous bone marrow adult mesenchymal stem cells expanded in vitro. Administered by Intrathecal injection (subarachnoid and intramedullary). Depending on centromedullary post-traumatic injury: bone marrow stromal stem cells administration (MSCs) at the minimum dose of 100x106 followed by subarachnoid administration of 30x106 MSCs,3 months later
  Mesenchymal stromal cell therapy
Arm/Group | Mesenchymal Stromal Cell Therapy
Number analyzed (Participants) | 12
Adverse events | 69

2. Secondary Outcome: Efficacy-Sensitivity Recovery Using ASIA Scale
Description: Sensitivity recovery was measured using the ASIA (American Spinal Injury Association) scale to measure the Surface sensitivity (LTS), pain sensitivity (PPS), and the degree of motor function in key muscles (MS). The sum of MS, LTS, and PPS configure total ASIA score. A minimum possible score is 0 points. A maximum possible score is 224 points for a patient with normal sensation.
  ASIA score was obtained before surgery, and 3, 6, 9 and 12 months after surgery. Mean and standard deviation for the 12 patients were obtained at all the time points and statistically analyzed.
Time Frame: sensitivity before surgery (baseline visit) and 3, 6, 9, 12 months after surgery (follow-up period)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mesenchymal Stromal Cell Therapy
Number analyzed (Participants) | 12
units on a scale
  Before Surgery | 165.92 (22.83)
  3 months after surgery | 181.25 (22.90)
  6 months after surgery | 189.83 (27.83)
  9 months after surgery | 200.75 (34.40)
  12 months after surgery | 213.25 (37.19)

3. Secondary Outcome: Efficacy-Changes in the Level of Chronic Pain Based on the IANR-SCIFRS Scale (Pain Section)
Description: Changes in the level of chronic pain, measured by the pain section of the IANR-SCIFRS (Spinal cord injury functional rating scale (SCI-FRS) of the international association of neuroestoratology (IANR). The minimum posible score is 0, and the máximum posible score is 48, being a score of 48 a normal functioning across all categories, and 0 a severe degree of functional hándicap (significant impact of daily life).
  Pain is classified as no pain; mild pain, ordinary pain killer, effective;severe pain, narcotics required; extreme pain, uncontrolled.
Time Frame: Changes in the level of Chronic pain before surgery (baseline visit) and 3, 6, 9, 12 months after surgery (follow-up period)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mesenchymal Stromal Cell Therapy
Number analyzed (Participants) | 12
units on a scale
  Before Surgery | 2.00 (0.95)
  3 months after surgery | 2.25 (0.97)
  6 months after surgery | 2.42 (0.90)
  9 months after surgery | 2.42 (0.90)
  12 months after surgery | 2.58 (0.79)

4. Secondary Outcome: Efficacy- Changes in the Neurophysiological Parameters Measured as the Number of Patients With SSEPs (Somatosensory Evoked Potentials)
Description: Changes in the neurophysiological parameters (SSEPs, somatosensory evoked potentials) measured as number of patients WITH SSEPs, each patient through underwent neurophysiological studies before treatment, as well as six and 12 months after surgery, paying attention mainly to the presence or abscence of somatosensory evoked potentials (SSEPs), the presence or absence of motor evoked potentials (MEPs) elicited by magnetic stimulation over the scalp, and to electromyographic (EMG) recording of motor unit potentials in infralesional muscles. Previous to cell therapy in any of the patients SSEPs were recorded.
Time Frame: Changes in the level neurophysiological parameters improvement (baseline visit) and 6, 12 months after surgery (follow-up period)
Measure: Number; unit: number of patients with SSEPs
Arm/Group | Mesenchymal Stromal Cell Therapy
Number analyzed (Participants) | 12
number of patients with SSEPs
  Before Surgery | 0
  6 months after surgery | 5
  12 months after surgery | 7

5. Secondary Outcome: Efficacy-Urodynamic Studies in Terms of máximum Cystometric Capacity
Description: Urodynamic studies in terms of voluntary micturition in flowmetry or in pressure/flow test, increase in bladder compliance. detrusor pressure (decrease on detrusor pressure is considered a clinical improvement). The neurogenic bladder is one of the biggest problems associated with SCI (spinal cord injury), with important personal and social implications.
Time Frame: Urodynamic studies before surgery and 12 months after surgery (follow-up period)
Measure: Mean (Standard Deviation); unit: cm/H2O
Arm/Group | Mesenchymal Stromal Cell Therapy
Number analyzed (Participants) | 12
cm/H2O
  Before Surgery | 77.50 (34.61)
  12 months after surgery | 54.58 (22.88)

6. Secondary Outcome: Efficacy-modification of Magnetic Resonance Imaging (MRI)
Description: Number of patients with a decrease in volume and hyperintensity of intramedullary lesions. In general, in the areas of SCI, variable degree of spinal cord atrophy and hiperintense images are observed. These images corresponds to cysts, gliosis and myelomalacia. After cell administration a reduction of supposed cyst and a decrease or disappearance of hyperintense lesions suggest a patient improvement.
Time Frame: changes in the spinal cord morphology on neuroimaging studies before surgery and 12 months after surgery (follow-up period)
Measure: Number; unit: Patients
Arm/Group | Mesenchymal Stromal Cell Therapy
Number analyzed (Participants) | 12
Patients
  Before Surgery | 0
  12 months after surgery | 7

ADVERSE EVENTS:
Time Frame: Along the study
Arm/Group | Mesenchymal Stromal Cell Therapy
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stromal Cell Therapy (N=12)
High level of cholesterol in blood (Metabolism and nutrition disorders) | 1 (1)
Pain (General disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
High level of alkaline phosphatase in blood (Metabolism and nutrition disorders) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 12 (24)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2)
Subcutaneous seroma (Injury, poisoning and procedural complications) | 1 (1)
Hemorrhoidectomy (Surgical and medical procedures) | 1 (1)
Pressure ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Intercostal nerualgia (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Saline extravasation (General disorders) | 1 (2)
Local edema (General disorders) | 1 (1)
Hyperthermia (General disorders) | 3 (5)
Thoracic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Urinary disconfort (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes